CLINICAL TRIAL: NCT06678763
Title: Combined Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy in Women With Inadvertently Morcellated Uterine Leiomyosarcoma: a Registry Study From a Tertiary Referral Hospital
Brief Title: Combined CRS With HIPEC in Women With Inadvertently Morcellated uLMS
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jing Li, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-939-01
Record Dates: First submitted 2024-11-03; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Uterine Leiomyosarcoma
Keywords: Cytoreductive surgery; Hyperthermic intraperitoneal chemotherapy; Morcellation; Uterine leiomyosarcoma;

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRS-HIPEC: The patient received open laparotomy cytoreduction surgery in the same principle as epithelial ovarian cancer surgery, and received intraperitoneal hyperthermic chemotherapy with docetaxel (75 mg/m²) and gemcitabine (1000 mg/m²) within 24 hours after surgery.
  Interventions: Procedure: CRS-HIPEC

INTERVENTIONS:
Procedure: CRS-HIPEC — Patients with uterine leiomyosarcoma who received unprotected morcellation were treated with cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy with docetaxel and gemcitabine.

SUMMARY:
For patients with benign tumors who undergo hysterectomy or myomectomy, minimally invasive gynecologic surgery (MIGS) has advantages over traditional laparotomy such as less trauma and faster recovery. The application of comminution technology is helpful for the implementation of MIGS. Uterine leiomyosarcoma (uLMS) is a malignant tumor that is difficult to diagnose preoperatively and is highly invasive. It is often diagnosed as a benign tumor before surgery. Occult uLMS will cause peritoneal dissemination after non-protective comminution surgery, leading to catastrophic outcomes and extremely poor prognosis. Hyperthermic intraperitoneal chemotherapy (HIPEC) is an important method for the treatment of peritoneal disseminated tumors and has been used in the treatment of gastrointestinal tumors and ovarian cancer. Recent studies have reported that it can significantly improve the progression-free survival (PFS) and overall survival (OS) rates of patients with recurrent uLMS and peritoneal metastasis. However, the efficacy and safety of this treatment for patients with accidental non-protective comminution of uLMS remain uncertain. This study will conduct a retrospective study to evaluate the efficacy and safety of CRS-HIPEC as the first-line treatment for accidentally morcellated uLMS.

DETAILED DESCRIPTION:
For patients undergoing hysterectomy or myomectomy for benign uterine tumors, minimally invasive gynecologic surgery (MIGS) has the advantages of fewer complications and faster recovery time compared with traditional laparotomy. Morcellation techniques, which are used to pulverize the uterus or myoma, facilitate the implementation of MIGS, especially for women with large uteruses or myomas or who are nulliparous. However, the safety of morcellation techniques has been controversial since the US Food and Drug Administration (FDA) issued a warning in 2014. The main concern is that unprotected morcellation may spread tissue fragments throughout the abdominal cavity. If a malignancy is present, such as uterine leiomyosarcoma (uLMS)-a highly invasive tumor that is difficult to diagnose preoperatively-this spread can have catastrophic consequences. The 5-year disease-specific survival rate for patients with uLMS who undergo unprotected morcellation is only 25.3%, while the 5-year disease-specific survival rate for patients who undergo complete tumor resection is 62.6%. Although the FDA recommends the use of tissue containment systems during laparoscopic morcellation, implementation of this recommendation varies worldwide, and endobag devices (tissue protection bags) are not universally available. Therefore, the management of peritoneal uLMS that disseminate after unprotected morcellation remains a major clinical challenge.

Hyperthermic intraperitoneal chemotherapy (HIPEC) is an important method for the treatment of peritoneal disseminated tumors. Cytoreductive surgery (CRS) combined with hyperthermic intraperitoneal chemotherapy (HIPEC) has shown efficacy in the treatment of peritoneal carcinomatosis in gastrointestinal and ovarian cancers. Recent studies have reported that it can significantly improve progression-free survival (PFS) and overall survival (OS) rates in patients with recurrent uLMS with peritoneal metastasis. A meta-analysis of 13 cases of recurrent uLMS conducted by Matsuzaki et al. in 2021 showed that the 3-year progression-free survival (PFS) and overall survival (OS) rates of patients who received CRS-HIPEC were 71.4% and 75.0%, respectively, compared with 0% and 50.1% for patients who received CRS alone. However, the efficacy and safety of this treatment for patients with accidentally comminuted uLMS remain uncertain.

In 2016, Sun Yat-sen Memorial Hospital of Sun Yat-sen University established a HIPEC program to routinely perform tumor reduction surgery and hyperthermic intraperitoneal chemotherapy (CRS-HIPEC) for patients with comminuted uLMS. Due to the limited availability of the HIPEC program outside our center, the HIPEC PROGRAM registry system was established to help refer patients from external institutions and receive CRS-HIPEC treatment. This study will conduct a retrospective study through the registration system, with patients who underwent unprotected morcellation surgery for occult uLMS and received CRS-HIPEC treatment as the research subjects, with progression-free survival (PFS) and overall survival (OS) as the primary outcomes, and the incidence of HIPEC-related ≥ grade 3 adverse events (AEs) as the secondary outcome, to evaluate the efficacy and safety of CRS-HIPEC as the first-line treatment for accidentally morcellated uLMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent myomectomy or hysterectomy for presumed benign disease and used non-protected morcellation and were subsequently pathologically diagnosed with uterine leiomyosarcoma.
* Patients underwent open laparotomy with similar surgical principles to epithelial ovarian cancer and achieved complete resection (R0 resection)
* Patients received closed hyperthermic intraperitoneal chemotherapy with docetaxel + gemcitabine after surgery.

Exclusion Criteria:

* Patients who received chemotherapy or radiotherapy previously.
* Incomplete follow-up data

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Patients with uterine leiomyosarcoma who received unprotected morcellation were treated with cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy with docetaxel and gemcitabine.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From completion of CRS-HIPEC to disease recurrence, assessed up to 120 months
  Time from completion of CRS-HIPEC to disease recurrence
Overall survival (OS) | From completion of CRS-HIPEC to death of any cause, assessed up to 120 months
  Time from completion of CRS-HIPEC to death of any cause

SECONDARY OUTCOMES:
Adverse Events (AE) | up to 3 weeks after CRS-HIPEC
  he adverse events would be graded according to Memorial Sloan-Kettering Cancer Center surgical secondary events (MSK SSE) grading system. The types and incidence of AEs will be recorded to evaluate the safety of CRS-HIPEC

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matsuzaki S, Matsuzaki S, Chang EJ, Yasukawa M, Roman LD, Matsuo K. Surgical and oncologic outcomes of hyperthermic intraperitoneal chemotherapy for uterine leiomyosarcoma: A systematic review of literature. Gynecol Oncol. 2021 Apr;161(1):70-77. doi: 10.1016/j.ygyno.2020.12.032. Epub 2021 Jan 6. PMID 33419612
- [Background] Xu X, Lin H, Wright JD, Gross CP, Boscoe FP, Hutchison LM, Schwartz PE, Desai VB. Association Between Power Morcellation and Mortality in Women With Unexpected Uterine Cancer Undergoing Hysterectomy or Myomectomy. J Clin Oncol. 2019 Dec 10;37(35):3412-3424. doi: 10.1200/JCO.19.00562. Epub 2019 Sep 16. PMID 31518176
- [Background] Graebe K, Garcia-Soto A, Aziz M, Valarezo V, Heller PB, Tchabo N, Tobias DH, Salamon C, Ramieri J, Dise C, Slomovitz BM. Incidental power morcellation of malignancy: a retrospective cohort study. Gynecol Oncol. 2015 Feb;136(2):274-7. doi: 10.1016/j.ygyno.2014.11.018. Epub 2014 Nov 26. PMID 25740603
- [Background] Senapati S, Tu FF, Magrina JF. Power morcellators: a review of current practice and assessment of risk. Am J Obstet Gynecol. 2015 Jan;212(1):18-23. doi: 10.1016/j.ajog.2014.07.046. Epub 2014 Jul 26. PMID 25072737
- [Background] Rayburn WF. Minimally Invasive Gynecologic Surgery: Improving Outcomes and Recovery While Reducing Discomfort and Cost. Obstet Gynecol Clin North Am. 2022 Jun;49(2):xiii-xiv. doi: 10.1016/j.ogc.2022.04.002. No abstract available. PMID 35636816